CLINICAL TRIAL: NCT07015697
Title: A Phase 1, Multicenter Trial of Subcutaneous Trastuzumab Deruxtecan in Participants With Metastatic Solid Tumors
Brief Title: A Study of Subcutaneous Trastuzumab Deruxtecan in Participants With Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-801
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Recurrent or Metastatic Solid Tumors
Keywords: T-DXd; solid tumor; subcutaneous
MeSH Terms: conditions — Recurrence | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Dose Escalation) (Experimental): Participants will receive Trastuzumab Deruxtecan subcutaneously at escalating doses. The recommended dose for expansion (RDE) will be calculated using data collected from this population.
  Interventions: Drug: Trastuzumab Deruxtecan
- Part 2 (Dose Expansion) (Experimental): Participants will receive Trastuzumab Deruxtecan subcutaneously at the recommended dose for expansion (RDE)
  Interventions: Drug: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — Dose Escalation Part: Trastuzumab Deruxtecan will be administered at escalating doses to determine the RDE.
  Expansion Part: Trastuzumab Deruxtecan will be administered at RDE.
  Other Names: T-DXd; ENHERTU®

SUMMARY:
This is a dose escalation, and dose expansion study of T-DXd plus hyaluronidase administered subcutaneously, to assess the safety, tolerability, PK and efficacy of SC T-DXd plus hyaluronidase in participants with metastatic solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Sign and date the ICF, prior to the start of any trial- specific qualification procedures.
2. Adults ≥18 years or the minimum legal adult age (whichever is greater).
3. a) Disease State: If HER2 status is required for eligibility (for all populations, except "Pan-tumor, heavily pretreated, with no SoC"), a documented HER2 test result must be available. A participant population would only be considered in regions where T-DXd is approved for that indication and an approved or validated test is available, if required per country regulations. Note: for all indications, all local HR testing and HER2 testing shall be per ASCO/CAP guidelines, as applicable, in the advanced setting, using a validated or approved test as required per local regulations. The most recent available samples should be used to confirm eligibility, if applicable. For full description of each population, see below. Breast Cancer: adults with pathologically documented unresectable or metastatic breast cancer HER2-positive BC: have received a prior anti-HER2-based regimen. For HER2-positive BC participants in Part 2 only, prior anti-HER2 based therapy should have been received in either:

   * the metastatic setting, or
   * the neoadjuvant or adjuvant setting and have developed disease recurrence during or within 6 months of completing therapy. HR-, HER2-low BC: have received a prior systemic cytotoxic therapy in the metastatic setting; or developed disease recurrence during or within 6 months of completing (neo)adjuvant chemotherapy. HR+, HER2-low/ultralow BC: have received previous ET AND an additional line of ET must not be the next line of treatment considered in the participant's best interest.
   * For participants in Part 2 with HR+ HER-2low/ultralow BC, the following criteria also apply:
   * had disease progression while receiving 1 previous line of ET with a CDK4/6i and is not expected to benefit from immediate use of a second line of ET, OR
   * had disease progression on at least 2 previous lines of ET with or without a target therapy such as CDK4/6, mTOR or PI3-K inhibitors) administered for the treatment of metastatic disease
   * of note:
   * If the 1 line was given while in the adjuvant setting, if disease recurrence occurred while on the first 24 months of adjuvant ET, that will be considered a line of therapy and only 1 additional line of ET will be required in the metastatic setting, with or without targeted therapy (such as CDK4/6, mTOR or PI3-K inhibitors)
   * Any progression after discontinuing or completing a course of adjuvant ET will not be considered a line of therapy
   * Single agent PARP inhibitor therapy does not count as ET or as cytotoxic is not considered a line of ET
   * Changes in dosing schedules, or discontinuations/restarting of the same drugs or the addition of a targeted therapy to an ET without progression (eg, adding a CDK4/6 inhibitor to a current aromatase inhibitor regimen) will not be considered separate lines of therapy.
   * participants may not have received more than 2 prior lines of cytotoxic therapy in the recurrent or metastatic setting. NSCLC, HER2 mut: adults with unresectable or metastatic NSCLC whose tumors have activating HER2 (ERBB2) mutations, and who have received a prior systemic therapy.

   Gastric Cancer, HER2-positive: adults with locally advanced or metastatic HER2-positive (IHC 3+ or IHC 2+/ISH+) gastric or gastroesophageal junction adenocarcinoma who have received a prior anti-HER2-based regimen Pan-tumor, HER2-positive: adults with unresectable or metastatic HER2-positive (IHC 3+) solid tumors who have received prior treatment or have no satisfactory alternative treatment options Heavily pretreated tumors: adults with unresectable or metastatic solid tumors (other than described above), who have received prior systemic treatment and have no satisfactory treatment alternative b) Part 2 only: At least 1 RECIST 1.1 measurable lesion on CT or MRI.
4. Radiologic or objective evidence of disease progression on or after the last systemic therapy prior to starting trial intervention.
5. Part 2 only: confirmation of availability of the most recent available adequate FFPE archival tumor tissue sample obtained in the advanced setting, or provision of newly obtained tumor tissue if clinically feasible and at an acceptable risk as determined by the Investigator.
6. ECOG PS of 0 to 1.

Key Exclusion Criteria:

1. Prior treatment with ADC that consists of an exatecan derivative that is a topoisomerase I inhibitor; NOTE exception for SDC 1 and 2, where prior exposure to such agents is permitted provided the following are met:

   1. At least 1 year has elapsed since last dose of exatecan derivative ADC.
   2. The participant did not discontinue nor reduce the dose due to toxicity.
   3. The participant did not experience any drug-related Grade 3/4 toxicity.
   4. The participant did not experience ILD of any grade while on or after the exatecan derivative ADC treatment.
2. Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug products.
3. Has a history of severe hypersensitivity reactions to other monoclonal antibodies.
4. Medical history of MI within 6 months before enrollment or symptomatic CHF (New York Heart Association class II to IV). Participants with troponin levels above ULN at screening (as defined by the manufacturer), and without any MI-related symptoms should have a cardiologic consultation during the Screening Period to rule out MI.
5. Has a corrected QT interval (QTcF) prolongation to > 480 ms (regardless of participant's sex) based on average of the screening triplicate 12-lead ECG.
6. Has a history of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing a Treatment Emergent Adverse Event (TEAE) | From the start of trial intervention to 21 days after the last dose, up to approximately 9 months
  TEAEs are defined as those Adverse Events (AEs) with start or worsening date during the on-treatment period (from the first dose date of trial intervention to 21 days after the last dose date of trial intervention).
Area Under Curve (AUC) | From the start of trial intervention to last dose, up to approximately 9 months
Number of Participants with Dose limiting toxicities (DLT) During the Dose-Escalation Phase | From the start of trial intervention to 21 days after the last dose, up to approximately 9 months

SECONDARY OUTCOMES:
Percentage of Participants with Anti-Drug Antibody (ADAs) | From baseline to post-baseline, up to approximately 12 months
Overall Response Rate (ORR) | From the enrollment/randomization date until documented disease progression, up to 12 months
  ORR is defined as the proportion of participants who achieved a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), as assessed by investigator per RECIST v1.1
Disease Control Rate (DCR) | From the enrollment/randomization date until documented disease progression, up to 12 months
  DCR is defined as the proportion of participants with a BOR of confirmed CR, confirmed PR, or stable disease (SD) per RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (6):
  - Research Site, Newport Beach, California
  - Research Site, Atlanta, Georgia
  - Research Site, Las Vegas, Nevada
  - Research Site, Charlotte, North Carolina
  - Research Site, Maumee, Ohio
  - Research Site, Nashville, Tennessee
- Japan (3):
  - Research Site, Chiba
  - Research Site, Kanagawa
  - Research Site, Tokyo
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
- Taiwan (3):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/